CLINICAL TRIAL: NCT02682316
Title: A Phase III Randomized Controlled Trial of Negative Pressure Wound Therapy in Post-Operative Incision Management
Brief Title: Negative Pressure Wound Therapy in Post-Operative Incision Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: 3M (Industry); Miami Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-309
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-01

CONDITIONS: Negative-Pressure Wound Therapy
Keywords: undergoing laparotomy; 15-309

ARMS (2):
- usual standard dry gauze used for wound management (Active Comparator): Patients who are randomized to the standard dry gauze arm will have the standard dry gauze placed at time of wound closure. Their dressing will be removed on post-operative day 2 as per routine departmental practice.
  Interventions: Other: dry gauze
- Prevena Negative Pressure Wound Therapy System (NPWT) (Experimental): Patients who are randomized to the Prevena Therapy System arm will have the Prevena Incision Management System device placed at time of wound closure. The device will be removed on day of discharge from the hospital or post-operative day 7, whichever comes first.
  Interventions: Device: The Prevena Incision Management System

INTERVENTIONS:
Other: dry gauze
  Arms: usual standard dry gauze used for wound management
Device: The Prevena Incision Management System
  Arms: Prevena Negative Pressure Wound Therapy System (NPWT)

SUMMARY:
The purpose of this study is to compare any good and bad effects of using the Prevena Incision Management System to using the usual standard dry gauze approach. The Prevena Incision Management System is a type of Negative Pressure Wound Therapy (NPWT). NPWT is a portable vacuum device made of a sponge-like foam that is applied over your incision to help draw fluid and debris out after surgery.

ELIGIBILITY:
Inclusion Criteria:

Criteria for Eligibility Prior to Surgery:

* Women of any BMI undergoing a laparotomy procedure for a presumed gynecologic malignancy, or morbidly obese (BMI ≥ 40) women undergoing a laparotomy for any indication
* or women who are morbidly obese (BMI>40) undergoing laparotomy for any indication
* Age ≥ 18

Criteria for Eligibility During Surgery:

* Women of any BMI undergoing a laparotomy procedure for a presumed gynecologic malignancy, or morbidly obese (BMI ≥ 40) women undergoing a laparotomy for any indication
* or women who are morbidly obese (BMI>40) undergoing laparotomy for any indication
* Age ≥ 18

Exclusion Criteria:

Exclusion prior to Surgery:

* Women undergoing panniculectomy at the time of laparotomy
* Women with sensitivity to silver

Exclusion during Surgery:

* Women with laparotomy incisions left open due to case classification as "contaminated" or "dirty"
* Women with laparotomy incisions unable to be closed primarily due to tissue or fascial damage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leitao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow-Up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow-Up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow-Up only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-Up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow-Up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville (Consent and Follow-Up only), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-Up only), Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- [Derived] Leitao MM Jr, Zhou QC, Schiavone MB, Cowan RA, Smith ES, Iasonos A, Veith M, Rafizadeh M, Curran K, Ramesh B, Chang K, Chi DS, Sonoda Y, Brown AK, Cosin JA, Abu-Rustum NR, Martino MA, Mueller JJ, Long Roche K, Jewell EL, Broach V, Lambrou NC, Diaz JP, Zivanovic O. Prophylactic Negative Pressure Wound Therapy After Laparotomy for Gynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2021 Feb 1;137(2):334-341. doi: 10.1097/AOG.0000000000004243. PMID 33416292
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Standard Dry Gauze Used for Wound Management: Patients who are randomized to the standard dry gauze arm will have the standard dry gauze placed at time of wound closure. Their dressing will be removed on post-operative day 2 as per routine departmental practice.
  dry gauze
- Prevena Negative Pressure Wound Therapy System (NPWT): Patients who are randomized to the Prevena Therapy System arm will have the Prevena Incision Management System device placed at time of wound closure. The device will be removed on day of discharge from the hospital or post-operative day 7, whichever comes first.
  The Prevena Incision Management System
Period: Overall Study
Arm/Group | Usual Standard Dry Gauze Used for Wound Management | Prevena Negative Pressure Wound Therapy System (NPWT)
Started | 294 | 289
Completed | 251 | 254
Not Completed | 43 | 35
Not completed — Benign Final Pathology | 27 | 26
Not completed — Reoperation before 30 days | 7 | 6
Not completed — Ineligible | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Standard Dry Gauze Used for Wound Management | Prevena Negative Pressure Wound Therapy System (NPWT) | Total
Number analyzed (Participants) | 294 | 289 | 583
Age, Continuous [Mean (Full Range); unit: years] | 60 [20 to 85] | 61 [18 to 66] | 60 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 289 | 583
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 22 | 38
  Not Hispanic or Latino | 278 | 267 | 545
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 23 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 23 | 37
  White | 245 | 233 | 478
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 10 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 294 | 289 | 583

OUTCOME MEASURES:

1. Primary Outcome: Number of Post-op Wound Complications
Description: Incidence of inpatient post-operative wound complications will be documented through the use of an inpatient data collection sheet. Incidence of outpatient post-operative wound complication will be documented through the use of an outpatient data collection sheet that will be completed by a provider at the time of the routine post-operative follow-up visit, which will occur at 30 days +/- 5 days after the day of surgery as well as through ongoing documentation of events as elicited through the institution's standard reporting system to collect information on enrolled patients.
Time Frame: 30 days +/- 5 days after surgery
Measure: Number; unit: Wound Complications
Arm/Group | Usual Standard Dry Gauze Used for Wound Management | Prevena Negative Pressure Wound Therapy System (NPWT)
Number analyzed (Participants) | 251 | 254
Wound Complications
  Inpatient wound complication | 2 | 5
  Outpatient wound complication | 42 | 36

ADVERSE EVENTS:
Time Frame: 30 days +/- 5 days after surgery
Arm/Group | Usual Standard Dry Gauze Used for Wound Management | Prevena Negative Pressure Wound Therapy System (NPWT)
All-Cause Mortality (participants affected / at risk) | 1/251 | 0/254
Serious Adverse Events (participants affected / at risk) | 51/251 | 69/254
Other Adverse Events (participants affected / at risk) | 11/251 | 44/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Standard Dry Gauze Used for Wound Management (N=251) | Prevena Negative Pressure Wound Therapy System (NPWT) (N=254)
Abdominal infection (Infections and infestations) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 4
Ascites (Gastrointestinal disorders) | 3 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Biliary fistula (Hepatobiliary disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Fever (General disorders) | 0 | 2
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 10 | 13
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Intraoperative splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Localized edema (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 2
Metabolism and nutrition disorders- Other, specify (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pain (General disorders) | 0 | 1
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 3
Ureteric anastomotic leak (Injury, poisoning and procedural complications) | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Standard Dry Gauze Used for Wound Management (N=251) | Prevena Negative Pressure Wound Therapy System (NPWT) (N=254)
Skin blistering (Skin and subcutaneous tissue disorders) | 3 | 33
Contact dermatitis (Skin and subcutaneous tissue disorders) | 4 | 6
Wound pain (Injury, poisoning and procedural complications) | 2 | 6
VAS pain level (Injury, poisoning and procedural complications) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT02682316/Prot_SAP_000.pdf